CLINICAL TRIAL: NCT02408861
Title: A Phase I Study of Ipilimumab and Nivolumab in Advanced HIV Associated Solid Tumors With Expansion Cohort in HIV Associated Solid Tumors and a Cohort of HIV-Associated Classical Hodgkin Lymphoma
Brief Title: Nivolumab and Ipilimumab in Treating Patients With HIV Associated Relapsed or Refractory Classical Hodgkin Lymphoma or Solid Tumors That Are Metastatic or Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00461; NCI-2015-00461 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PAMC-095_R03PAPP01; AMC-095; AMC-095 (Other: AIDS Malignancy Consortium); AMC-095 (Other: CTEP); U01CA121947 (NIH); UM1CA121947 (NIH)
Record Dates: First submitted 2015-04-03; First posted 2015-04-06 (Estimated); Results first posted 2025-09-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Solid Neoplasm; Anal Carcinoma; HIV Infection; Kaposi Sarcoma; Lung Carcinoma; Metastatic Malignant Solid Neoplasm; Recurrent Classic Hodgkin Lymphoma; Refractory Classic Hodgkin Lymphoma; Unresectable Solid Neoplasm; HIV-associated Cancers
Keywords: Immunotherapy; Immune check point blockade; Anti-CTLA-4 antibody; Anti-PD1 antibody; Phase 1; Dose de-escalation; Dose expansion
MeSH Terms: conditions — Anus Neoplasms; HIV Infections; Sarcoma, Kaposi; Lung Neoplasms; Neoplasm Metastasis | interventions — Specimen Handling; Biopsy; Ipilimumab; CTLA-4 Antigen; Nivolumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Dose De-escalation Single Agent Nivolumab Stratum 1 (Experimental): Stratum 1 will enroll participants with T lymphocyte CD4+ count above 200/mm3. Stratum 1 dosing will start with a full dose of nivolumab 3 mg/kg (dose level 1) and one dose de-escalation is allowed; after evaluating dosing for single agent nivolumab. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Nivolumab
- Dose De-escalation Single Agent Nivolumab Stratum 2 (Experimental): Stratum 2 will enroll participants with T lymphocyte CD4+ count between 100 to 200/mm3.
  Stratum 2 will start enrolling after completion of stratum 2 dose deescalation. The dosing will begin at the single-agent therapy MTD for Stratum 1 (dose level 1 or -1). Stratum 2 will not be allowed to escalate beyond the MTD for Stratum 1. Only 1 dose de-escalation will be allowed.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Nivolumab
- Dose De-escalation Cohort Combination Therapy (Nivolumab and Ipilimumab) Stratum 1 (Experimental): Stratum 1 dosing will start with a full dose of nivolumab 3 mg/kg (dose level 1) and one dose de-escalation is allowed; Participants will be treated with 240 mg of nivolumab and 1 mg/kg of ipilimumab will be added to evaluate combination therapy (dose level 2) with one dose de- escalation allowed. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Biological: Nivolumab
- Dose De-escalation Cohort Combination Therapy (Nivolumab and Ipilimumab) Stratum 2 (Experimental): Stratum 2 will enroll participants with lymphocyte T CD4+ count between 100-200/mm3 Participants will be treated with 240 mg of nivolumab and 1 mg/kg of ipilimumab will be added to evaluate combination therapy (dose level 2) with one dose de- escalation allowed. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Biological: Nivolumab
- Solid Tumors Dose Expansion Cohort Single Agent Nivolumab (Experimental): Participants with incurable solid tumors will be treated at single agent nivolumab 240 mg every 2 weeks. Only those histologies that are not known to respond to single agent nivolumab will be excluded (i.e., pancreas, prostate, MSS colorectal cancer, unless results from another clinical trial showing non-response in another tumor type become available in the future). Up to 24 participants will be enrolled.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Nivolumab
- Combination Regimen Expansion Cohort (Experimental): The combination therapy at MTD of Nivolumab and Ipilimumab regimen will be studied in a dose expansion cohort (up to 12 participants) limited to only participants with Kaposi sarcoma, lung cancer, and anal cancer.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Biological: Nivolumab
- Classical Hodgkin Lymphoma Cohort (Experimental): Single agent Nivolumab therapy at MTD dose from dose-de-escalation will be administered in participants with classical Hodgkin's Lymphoma with a fixed dose of 240 mg q 2 week.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Biological: Nivolumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
  Arms: Classical Hodgkin Lymphoma Cohort
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Combination Regimen Expansion Cohort; Dose De-escalation Cohort Combination Therapy (Nivolumab and Ipilimumab) Stratum 1; Dose De-escalation Cohort Combination Therapy (Nivolumab and Ipilimumab) Stratum 2
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
  Arms: Classical Hodgkin Lymphoma Cohort

SUMMARY:
This phase I trial studies the side effects and best dose of nivolumab when given with ipilimumab in treating patients with human immunodeficiency virus (HIV) associated classical Hodgkin lymphoma that has returned after a period of improvement (relapsed) or does not respond to treatment (refractory), or solid tumors that have spread from where it first started to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ipilimumab is an antibody that acts against a molecule called cytotoxic T-lymphocyte antigen 4 (CTLA-4). CTLA-4 controls a part of the immune system by shutting it down. Nivolumab is a type of antibody that is specific for human programmed cell death 1 (PD-1), a protein that is responsible for destruction of immune cells. Giving ipilimumab with nivolumab may work better in treating patients with HIV associated classical Hodgkin lymphoma or solid tumors compared to ipilimumab with nivolumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate safety and feasibility of ipilimumab and nivolumab at the standard doses of drug in solid tumor and relapsed refractory HIV-classical Hodgkin lymphoma (cHL) participants with human immunodeficiency virus (HIV) infection given the possibility of increased toxicity based on immune activation, co-morbidity, or interference with highly active antiretroviral therapy (HAART) therapy. (Dose De-escalation and Dose Expansion Cohorts)

SECONDARY OBJECTIVES:

I. To evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab, on immune function (HIV viral load in plasma using conventional assay, CD4+ and CD8+ cells). (Dose De-escalation Cohort) II. To preliminarily assess objective response rates associated with treatment for commonly represented solid tumors (Kaposi sarcoma, anal cancer, and lung cancer) and relapsed refractory HIV-cHL. (Solid Tumor Dose Expansion and cHL Cohorts) III. To evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab, on immune function (HIV viral load in plasma using conventional HIV assay, CD4+, and CD8+ cells). (Solid Tumor Dose Expansion and cHL Cohorts)

EXPLORATORY OBJECTIVES:

I. Understand the immune response to agent in the context of antiretroviral therapy (ART), of altered immune function, and repertoire due to prior HIV infection.

Ia. To evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab, on intratumor immune cells by immunohistochemistry (IHC) such as PD1, programmed cell death 1 ligand 1 (PDL-1), and others.

Ib. To evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab on circulating cytokine markers by multiplex assay, such as: interleukin (IL)-2, IL-4, IL-6, IL-10, IL-8, interferon gamma-induced protein 10 (IP10), chemokine (C-X-C motif) ligand 13 (CXCL13), interferon (IFN)-gamma, tumor necrosis factor (TNF)-alpha, soluble IL-2 receptor (sIL2R)-alpha, sCD27, soluble TNF receptor (sTNFR)1, and sTNFR2.

II. To understand the response of human tumor viruses (human papillomavirus [HPV], Epstein-Barr virus [EBV], Kaposi's sarcoma-associated herpesvirus [KSHV]) to agent.

IIa. To evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab on herpesvirus loads (EBV, KSHV, cytomegalovirus [CMV]) in plasma.

IIb. To evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab on latent herpesvirus (EBV, KSHV, CMV) in peripheral blood mononuclear cells (PBMC).

IIc. To evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab on herpesvirus specific CD8 and CD4 T cells in PBMC.

IId. In cases of Kaposi sarcoma, to evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab on viral transcription in tumor biopsies.

IIe. In cases of anal cancer, to evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab on HPV types in anal swabs, when feasible.

III. Understand the response of HIV to agent. IIIa. To evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab on latent HIV loads in PBMC using outgrowth assay.

IIIb. To evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab on HIV reactive T cells.

OUTLINE: This is a dose-escalation study of nivolumab.

Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Patients in dose level 2 also receive ipilimumab IV over 90 minutes on day 1 of every third cycle of nivolumab, and patients in dose level -2 also receive ipilimumab IV over 90 minutes on day 1 of every sixth cycle of nivolumab. Treatment repeats every 14 days for up to 46 cycles of nivolumab (with ipilimumab if receiving dose level 2 or -2) in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study. Patients undergo positron emission tomography (PET) and computed tomography (CT) during screening and on study. Patients undergo bone marrow biopsy on screening and may undergo it during follow up.

After completion of study treatment, patients are followed up for 16 weeks or 112 days (based on 5 half lives).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed solid tumor malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; participants with uncontrolled Kaposi sarcoma are permitted (KS must be increasing despite HAART and HIV suppression for greater than or equal to 2 months, or stable KS despite HAART for greater than or equal to 3 months)

  * For participants in the 24 participant solid tumor cohort, only those histologies not known to respond to single agent nivolumab (such as pancreas, prostate, and microsatellite stable [MSS] colorectal cancer) will be excluded
  * For participants in the relapsed refractory HIV-cHL expansion cohort, participants must have histologically confirmed, relapsed/refractory (defined as relapsed/refractory to one or greater lines of therapy) HIV-associated classical Hodgkin lymphoma
* HIV-1 infection, as documented by any federally approved, licensed HIV rapid test performed in conjunction with screening (or enzyme linked immunosorbent assay [ELISA], test kit, and confirmed by Western blot or other approved test); alternatively, this documentation may include a record demonstrating that another physician has documented the participant's HIV status based on either: 1) approved diagnostic tests, or 2) the referring physician's written record that HIV infection was documented, with supporting information on the participant's relevant medical history and/or current management of HIV infection
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam; scans must have been performed within 4 weeks prior to registration; Note: for participants with Kaposi sarcoma, the following apply: at least five measurable cutaneous KS lesions or any number of lesions with systemic unresectable disease with no previous local radiation, surgical, or intralesional cytotoxic therapy that would prevent response assessment
* Prior therapy for metastatic disease permitted; at least 4 weeks must have elapsed since prior chemotherapy or biological therapy, 6 weeks if the regimen included carmustine (BCNU) or mitomycin C; radiotherapy must be completed at least 4 weeks prior to registration
* Age > 18 years, because no dosing or AE data are currently available on the use of ipilimumab in combination with nivolumab in participants <18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* PARTICIPANTS NOT ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Leukocytes >= 2,000/mm^3 (within 2 weeks prior to enrollment)
* PARTICIPANTS NOT ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Absolute neutrophil count >= 1,000/mm^3 (within 2 weeks prior to enrollment)
* PARTICIPANTS NOT ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Platelets >= 75,000/mm^3 (within 2 weeks prior to enrollment)
* PARTICIPANTS NOT ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) =< 3 x ULN for subjects with Gilbert's disease or with atazanavir- or indinavir-induced unconjugated hyperbilirubinemia without aspartate aminotransferase (AST) or alanine aminotransferase (ALT) elevation and must have a total bilirubin less than 3.0 mg/dL (within 2 weeks prior to enrollment)
* PARTICIPANTS NOT ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Serum lipase and amylase < 1.5 x ULN (within 2 weeks prior to enrollment)
* PARTICIPANTS NOT ON THE HODGKIN LYMPHOMA EXPANSION COHORT: AST (serum glutamic oxaloacetic transaminase [SGOT])/ALT (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN (within 2 weeks prior to enrollment)
* PARTICIPANTS NOT ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Creatinine < 1.5 UNL or creatinine clearance (CrCl) > 50 ml/min (within 2 weeks prior to enrollment)
* PARTICIPANTS NOT ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Hemoglobin >= 9 g/dL (within 2 weeks prior to enrollment)
* PARTICIPANTS NOT ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Serum albumin >= 2.8 g/dL (within 2 weeks prior to enrollment)
* PARTICIPANTS ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Leukocyte count: no lower limit (within 2 weeks prior to enrollment) (participants may receive granulocyte colony stimulating factor [GCSF] and transfusions to meet these parameters)
* PARTICIPANTS ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Absolute neutrophil count: >= 1,000/mm^3, unless decreased due to bone marrow involvement with lymphoma (within 2 weeks prior to enrollment) (participants may receive GCSF and transfusions to meet these parameters)
* PARTICIPANTS ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Platelets: >= 75,000/mm^3, unless decreased due to bone marrow involvement with lymphoma (within 2 weeks prior to enrollment) (participants may receive GCSF and transfusions to meet these parameters)
* PARTICIPANTS ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Hemoglobin: >= 9 g/dL unless bone marrow involvement secondary to Hodgkin lymphoma is present (within 2 weeks prior to enrollment) (participants may receive GCSF and transfusions to meet these parameters)
* PARTICIPANTS ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Total bilirubin: =< 1.5 x institutional upper limit of normal (ULN), or =< 3 x ULN for participants with Gilbert's disease or with atazanavir- or indinavir-induced unconjugated hyperbilirubinemia without AST or ALT elevation, and must have a total bilirubin less than 3.0 mg/dL) (within 2 weeks prior to enrollment) (participants may receive GCSF and transfusions to meet these parameters)
* PARTICIPANTS ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Serum lipase and amylase < 1.5 x ULN (within 2 weeks prior to enrollment) (participants may receive GCSF and transfusions to meet these parameters)
* PARTICIPANTS ON THE HODGKIN LYMPHOMA EXPANSION COHORT: AST (SGOT)/ALT (SGPT): =< 3 x ULN (within 2 weeks prior to enrollment) (participants may receive GCSF and transfusions to meet these parameters)
* PARTICIPANTS ON THE HODGKIN LYMPHOMA EXPANSION COHORT: Creatinine: < 1.5 x upper normal limit (UNL) or CrCl > 50ml/min (within 2 weeks prior to enrollment) (participants may receive GCSF and transfusions to meet these parameters)
* HIV viral load should be well suppressed, defined as below the limit of detection of the local assay or below 75 copies/mL by Food and Drug Administration (FDA)-approved assays, within 4 weeks prior to registration
* CD4 counts:

  * For Stratum 1: CD4+ cell count greater than 200 cells/mm^3 obtained within 2 weeks prior to enrollment at any United States (U.S.) laboratory that has a clinical laboratory improvement amendments (CLIA) certification or its equivalent
  * For Stratum 2: CD4 cell count between 100-200 cells/mm^3 obtained within 2 weeks prior to enrollment at any U.S. laboratory that has a clinical laboratory improvement amendments (CLIA) certification or its equivalent
  * Expansion Cohort: CD4 cell count for this cohort will be specified once Stratum 1 and Stratum 2 have completed enrollment
  * Solid Tumor Expansion Cohort: CD4+ cell count greater than 200 cells/mm^3 obtained within 2 weeks prior to enrollment at any U.S. laboratory that has a clinical laboratory improvement amendments (CLIA) certification or its equivalent
  * cHL Cohort: CD4 cell count of at least 100 cells/mm^3
* Participants must be purified protein derivative (PPD) negative; alternatively, the QuantiFERON-tuberculosis (TB) Gold In-Tube (QFT-GIT) assay can be used; an individual is considered positive for M. tuberculosis infection if the IFN-gamma response to TB antigens is above the test cut-off (after subtracting the background IFN-gamma response in the negative control); the result must be obtained within 12 weeks prior to enrollment; PPD positive (or Quantiferon assay positive) participants are permitted if prophylaxis has been completed prior to enrollment
* The effects of nivolumab and ipilimumab on the developing human fetus are unknown; for this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of childbearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; WOCBP should use an adequate method to avoid pregnancy for 6 months after the last dose of investigational drug; women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropic [HCG]) within 72 hours prior enrollment and the start of nivolumab; women must not be breastfeeding; men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception; WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 6 months after the last dose of investigational product; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately
* Participants MUST receive appropriate care and treatment for HIV infection, including antiretroviral medications when clinically indicated, and should be under the care of a physician experienced in HIV management; participants will be eligible regardless of antiretroviral medication (including no antiretroviral medication) provided there is no intention to initiate therapy or the regimen has been stable for at least 4 weeks with no intention to change the regimen within 12 weeks following enrollment
* Participants who have hepatitis C (both reactive anti-hepatitis C virus [HCV] antibody and detectable HCV ribonucleic acid [RNA]) and hepatitis B (hepatitis B surface antigen [HBsAg] positive and anti-hepatitis B core [HBc]-total positive), may be enrolled, provided total bilirubin is =< 1.5 x institutional ULN, and AST (SGOT) and ALT (SGPT) must be =< 3 X institutional upper limit of normal, and hepatitis B virus (HBV) deoxyribonucleic acid (DNA) < 100 IU/mL (if hepatitis B positive) within 2 weeks prior to enrollment
* Ability to understand and to sign a written informed consent document
* Criteria for Solid Tumor Expansion and Lymphoma Cohorts:

  * Inclusion and exclusion criteria for this cohort are the same as above, with the following rule for CD4 count based on tolerability in Phase I; if, participants with lymphocyte T CD4 count between 100-200/mm^3 (Stratum 2) are shown to tolerate treatment in the Phase I dose de-escalation portion at the same dose level as those with CD4 counts > 200/mm^3 (Stratum 1), participants in the expansion cohort with CD4 counts >= 100/mm^3 are permitted; otherwise, the expansion is open to all solid tumor patients except those whose tumors are known not to respond to nivolumab (pancreas, prostate and MSS colon cancer); for the relapsed refractory HIV-cHL cohort, participants with CD4 count >= 100/mm^3 are permitted

Exclusion Criteria:

* Participants who have received any other investigational agents within the 4 weeks prior to enrollment; concurrent radiation therapy is not permitted, except palliative (limited-field) radiation therapy, if all of the following criteria are met:

  * Repeat imaging demonstrates no new sites of bone metastases
  * The lesion being considered for palliative radiation is not a target lesion
* Participants with known brain metastases or leptomeningeal metastases must be excluded unless they qualify for enrollment as described below because of poor prognosis and concerns regarding progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; participants with brain metastases are permitted if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks or more after treatment is complete and within 4 weeks prior to the first dose of nivolumab administration
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ipilimumab, nivolumab, or other agents used in study, or history of severe hypersensitivity reaction to any monoclonal antibody
* Participants should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 2 weeks of study drug administration; these drugs may interfere with the activity of ipilimumab and nivolumab if administered at the time of the first ipilimumab dose; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; participants are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if >= 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted; use of anabolic steroids is permitted
* Participants with clinical or radiographic evidence of pancreatitis are excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Participants should be excluded if they have had prior treatment with an anti-PD-1, anti-programmed cell death ligand 1 (PD-L1), anti-programmed cell death ligand 2 (PD-L2), anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways; prior immune modulating therapy including vaccines may be eligible; prior immune events must be evaluated and the risk for new events which may represent continued sub clinical disease or a new process at previously damaged site or immune potentiation (e.g. ipilimumab followed by IL2 causing bowel perforation, ipilimumab followed by indoleamine 2,3-dioxygenase [IDO] inhibitor resulting in clinical hypophysitis); please keep in mind that inflammatory events may occur weeks to months following the last dose of ipilimumab and possibly nivolumab; assessment of potential effects of prior therapy should include:

  * Immune status
  * Organ damage
  * Risk of autoimmunity
  * Immunopotentiation
* The participant has not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 from toxicity due to all prior therapies except =< grade 2 alopecia, neuropathy, and other non-clinically significant adverse events (AEs)
* The participant has a primary brain tumor
* Participant has >= grade 2 diarrhea (participants with grade 1 diarrhea are eligible provided stool for ova/parasites and stool cryptosporidium studies are negative)
* Opportunistic infection within the last 3 months
* Participants with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and participants with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease; participants with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; participants with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and participants with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible; participants are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Participants who have had evidence of Clostridium (C.) difficile infection, active or acute diverticulitis, intra-abdominal abscess, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis, which are known risk factors for bowel perforation, should be evaluated for the potential need for additional treatment before coming on study
* cHL COHORT ONLY: history of allogeneic transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Rajdev, Principal Investigator — AIDS Malignancy Consortium
Locations (34):
- United States (32):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Center for Clinical AIDS Research and Education, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - FHCC South Lake Union, Seattle, Washington
- Australia (2):
  - Saint Vincent's Hospital, Darlinghurst, New South Wales
  - University of New South Wales, Sydney, New South Wales

REFERENCES:
- [Derived] Rajdev L, Jackie Wang CC, Joshi H, Lensing S, Lee J, Ramos JC, Baiocchi R, Ratner L, Rubinstein PG, Ambinder R, Henry D, Streicher H, Little RF, Chiao E, Dittmer DP, Einstein MH, Cesarman E, Mitsuyasu R, Sparano JA; AIDS Malignancy Consortium. Assessment of the safety of nivolumab in people living with HIV with advanced cancer on antiretroviral therapy: the AIDS Malignancy Consortium 095 Study. Cancer. 2024 Mar 15;130(6):985-994. doi: 10.1002/cncr.35110. Epub 2023 Nov 14. PMID 37962072
- [Derived] Rasmussen TA, Rajdev L, Rhodes A, Dantanarayana A, Tennakoon S, Chea S, Spelman T, Lensing S, Rutishauser R, Bakkour S, Busch M, Siliciano JD, Siliciano RF, Einstein MH, Dittmer DP, Chiao E, Deeks SG, Durand C, Lewin SR. Impact of Anti-PD-1 and Anti-CTLA-4 on the Human Immunodeficiency Virus (HIV) Reservoir in People Living With HIV With Cancer on Antiretroviral Therapy: The AIDS Malignancy Consortium 095 Study. Clin Infect Dis. 2021 Oct 5;73(7):e1973-e1981. doi: 10.1093/cid/ciaa1530. PMID 33677480

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started in October 2015 and ended June 2023 across 7 different cohorts, and 17 study sites.
Pre-assignment Details: Participants with histologically confirmed solid malignancy and HIV infection. Solid malignancy must be metastatic or unresectable and standard curative or palliative measures are nonexistent or no longer effective. Uncontrolled Kaposi sarcoma is permitted. Participants with relapsed refractory HIV-associated classical Hodgkin lymphoma (HIV-cHL) as a separate cohort.
Groups:
- Dose De-escalation Nivolumab 3mg/kg (Stratum 1): Nivolumab 3 mg/kg body weight (Dose level 1) Stratum 1: Participants with CD4+ count > 200/mm3.
  Start with a full dose of nivolumab 3 mg/kg (dose level 1) and one dose de-escalation is allowed; after evaluating dosing for single agent nivolumab then participants will be treated with 240 mg of nivolumab. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
- Dose De-escalation Nivolumab 3 mg/kg (Stratum 2): Nivolumab 3 mg/kg body weight (Dose level 1) Stratum 2 : Participants with CD4+ count between 100-200/mm3.
  Enrollment Stratum 2 will begin after Stratum 1 has completed.
  Stratum 2 dosing will begin at the single-agent therapy MTD for Stratum 1 (dose level 1 or -1). Stratum 2 will not be allowed to escalate beyond the MTD for Stratum 1. Only 1 dose de-escalation will be allowed.
- Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1): Nivolumab 240mg and Ipilimumab 1 mg/kg (Dose level 2); Stratum 1: CD4 count >200 per mm3;
  No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
- Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2): Nivolumab 240 mg and Ipilimumab 1mg/kg (Dose level 2); Stratum 2: participants with lymphocyte T CD4+ count between 100-200/mm3;
  Participants will be treated with 240 mg of nivolumab and 1 mg/kg of ipilimumab will be added to evaluate combination therapy (dose level 2) with one dose de- escalation allowed. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
- Dose Expansion Nivolumab 240 mg q2w in Solid Tumors: Participants with incurable solid tumors will be treated at single agent nivolumab 240 mg every 2 weeks. Only those histologies that are not known to respond to single agent nivolumab will be excluded (i.e., pancreas, prostate, MSS colorectal cancer, unless results from another clinical trial showing non-response in another tumor type become available in the future). Up to 24 participants will be enrolled.
- Dose Expansion Nivolumab 240 mg q2w and Ipilimumab 1 mg/kg q6w: The combination therapy MTD will be studied in a dose expansion cohort (up to 12 participants) limited to only participants with Kaposi sarcoma, lung cancer, and anal cancer.
- Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma: Single agent Nivolumab therapy will be administered in participants with classical Hodgkin's Lymphoma with a fixed dose of 240 mg q 2 week.
Period: Overall Study
Arm/Group | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors | Dose Expansion Nivolumab 240 mg q2w and Ipilimumab 1 mg/kg q6w | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma
Started | 6 | 9 | 7 | 4 | 24 | 20 | 9
Number of DLTs experienced within 6 weeks | 0 | 0 | 1 | 0 | 0 (DLT not evaluated for this cohort) | 0 (DLT not evaluated for this cohort) | 0 (DLT not evaluated for this cohort)
Patients receiving de-escalated dose of Nivolumab (1 mg/kg) | 0 | 0 | 0 | 0 | 0 (De-escalation Not Applicable) | 0 (De-escalation Not Applicable) | 0 (De-escalation Not Applicable)
Completed | 3 | 5 | 2 | 1 | 10 | 13 | 6
Not Completed | 3 | 4 | 5 | 3 | 14 | 7 | 3
Not completed — Death | 0 | 3 | 1 | 2 | 4 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 4 | 2 | 1
Not completed — Disease Progression | 0 | 0 | 1 | 0 | 3 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other Treatment | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dose De-escalation Nivolumab 3mg/kg (Stratum 1): Stratum 1 will enroll participants with CD4+ count above 200/mm3. Start with a full dose of nivolumab 3 mg/kg (dose level 1) and one dose de-escalation is allowed; after evaluating dosing for single agent nivolumab then participants will be treated with 240 mg of nivolumab. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
- Dose De-escalation Nivolumab 3 mg/kg (Stratum 2): Stratum 2 will enroll participants with CD4+ count between 100-200/mm3. Enrollment in Stratum 2 will begin after Stratum 1 has completed. Stratum 2 dosing will begin at the single-agent therapy MTD for Stratum 1 (dose level 1 or -1). Stratum 2 will not be allowed to escalate beyond the MTD for Stratum 1. Only 1 dose de-escalation will be allowed.
- Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1): Stratum 1 will enroll participants with CD4+ count above 200/mm3. Participants will be treated with 240 mg of nivolumab and 1 mg/kg of ipilimumab will be added to evaluate combination therapy (dose level 2) with one dose de- escalation allowed. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
- Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2): Stratum 2 will enroll participants with lymphocyte T CD4+ count between 100-200/mm3.
  Participants will be treated with 240 mg of nivolumab and 1 mg/kg of ipilimumab will be added to evaluate combination therapy (dose level 2) with one dose de- escalation allowed. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
- Total: Total of all reporting groups
Arm/Group | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors | Dose Expansion Nivolumab 240 mg q2w and Ipilimumab 1 mg/kg q6w | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma | Total
Number analyzed (Participants) | 6 | 9 | 7 | 4 | 24 | 20 | 9 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (6.2) | 59.4 (4.3) | 57.0 (6.6) | 45.8 (16.8) | 49.6 (11.2) | 52.6 (17.0) | 46.1 (9.8) | 51.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 0 | 3 | 1 | 0 | 7
  Male | 5 | 9 | 5 | 4 | 21 | 19 | 9 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 0 | 3 | 4 | 3 | 13
  Not Hispanic or Latino | 6 | 8 | 5 | 4 | 19 | 15 | 6 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 4 | 7 | 6 | 1 | 23
  White | 4 | 6 | 4 | 0 | 16 | 12 | 8 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 5
ECOG Grade of Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status, is a standardized scale used to assess how well a cancer patient performs daily activities. It helps to determine the extent of a patient's physical function and ability to tolerate treatment.
  ECOG 0 are fully active, able to carry out all activities without restriction. ECOG 1 indicates patients perceive restricted in strenuous physical activity, but ambulatory and able to carry out light or sedentary work.
  Patients with ECOG >=2 were excluded in this study. The ECOG grades are described at https://ecog-acrin.org/
  Participants
    ECOG Grade 0 | 3 | 2 | 2 | 1 | 11 | 10 | 4 | 33
    ECOG Grade 1 | 3 | 7 | 5 | 3 | 13 | 10 | 5 | 46
Count by cancer type [Count of Participants; unit: Participants]
  Kaposi's Sarcoma | 0 | 0 | 2 | 1 | 15 | 15 | 0 | 33
  Hodgkin's lymphoma | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9
  Anal Cancer | 0 | 5 | 0 | 1 | 1 | 2 | 0 | 9
  Lung cancer | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 6
  Colon cancer | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 4
  Head and Neck Cancer | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  Other cancer types | 4 | 1 | 2 | 2 | 5 | 1 | 0 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Nivolumab
Description: Will be defined as the starting dose level at which 1/6 subjects experience dose limiting toxicity (DLT) with the next higher dose having at least >= 2 participants encountering DLT. Toxicity data will be presented by type and severity for each dose group and overall; the incidence of toxicity related dose reductions and treatment discontinuations will be summarized.
Time Frame: Each patient will be evaluated for DLT for the safety evaluation period of 6 weeks
Population: Safety evaluable population treated with at least a single dose of Nivolumab.
Measure: Number; unit: mg/kg
Groups:
- Dose De-escalation Nivolumab 3 mg/kg (Stratum 1): Stratum 1 will enroll participants with CD4+ count above 200/mm3. Start with a full dose of nivolumab 3 mg/kg (dose level 1) and one dose de-escalation is allowed; after evaluating dosing for single agent nivolumab then participants will be treated with 240 mg of nivolumab. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
Arm/Group | Dose De-escalation Nivolumab 3 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2)
Number analyzed (Participants) | 6 | 9
mg/kg | 3 | 3

2. Primary Outcome: Dose Limiting Toxicities (DLTs) Observed in Dose De-escalation Cohorts
Description: Incidence of DLTs during the safety evaluation period of 6 weeks at a given dose from the first dose of treatment.
Time Frame: 6 weeks from the first dose of Nivolumab
Population: Patients evaluated for safety during 6 weeks from the first dose
Measure: Count of Participants; unit: Participants
Groups:
- Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 1): Stratum 1 dosing will start with a full dose of nivolumab 3 mg/kg (dose level 1) and one dose de-escalation is allowed;
  Participants will be treated with 240 mg of nivolumab and 1 mg/kg of ipilimumab will be added to evaluate combination therapy (dose level 2) with one dose de- escalation allowed. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
- Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2): Stratum 2 will enroll participants with lymphocyte T CD4+ count between 100-200/mm3
  Participants will be treated with 240 mg of nivolumab and 1 mg/kg of ipilimumab will be added to evaluate combination therapy (dose level 2) with one dose de- escalation allowed. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
Arm/Group | Dose De-escalation Nivolumab 3 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 1) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2)
Number analyzed (Participants) | 6 | 9 | 7 | 4
Participants | 0 | 0 | 1 | 0

3. Primary Outcome: Incidence of Adverse Events According to NCI CTCAE v5.0
Description: Number of adverse events that are either possibly, probably or definitely attributed to study intervention.
  In case an adverse event as per the CTCAE v5.0 occurs within a same patient, an instance with the highest severity of the adverse event is counted. Separate event-instances are reported otherwise.
Time Frame: Participants will be followed for 16 weeks or 112 days after removal from study treatment, or until death, whichever occurs first.
Measure: Number; unit: Events
Groups:
- Dose De-escalation Nivolumab 3mg/kg (Stratum 2): Nivolumab 3 mg/kg body weight (Dose level 1) Stratum 2 : Participants with CD4+ count between 100-200/mm3.
  Enrollment Stratum 2 will begin after Stratum 1 has completed.
  Stratum 2 dosing will begin at the single-agent therapy MTD for Stratum 1 (dose level 1 or -1). Stratum 2 will not be allowed to escalate beyond the MTD for Stratum 1. Only 1 dose de-escalation will be allowed.
- Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 2): Nivolumab 240 mg and Ipilimumab 1mg/kg (Dose level 2); Stratum 2: participants with lymphocyte T CD4+ count between 100-200/mm3;
  Participants will be treated with 240 mg of nivolumab and 1 mg/kg of ipilimumab will be added to evaluate combination therapy (dose level 2) with one dose de- escalation allowed. No intra-participant dose escalations will be allowed. The safety evaluation period is 6 weeks at a given dose level.
- Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg: The combination therapy MTD will be studied in a dose expansion cohort (up to 12 participants) limited to only participants with Kaposi sarcoma, lung cancer, and anal cancer.
Arm/Group | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3mg/kg (Stratum 2) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 2) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors | Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma
Number analyzed (Participants) | 6 | 9 | 7 | 4 | 24 | 20 | 9
Events
  Adverse Events | 27 | 29 | 26 | 8 | 54 | 72 | 29
  Serious Adverse Events | 3 | 5 | 2 | 1 | 5 | 3 | 2

4. Secondary Outcome: Objective Response Rate
Description: The proportion of patients achieving objective responses (by Response Evaluation Criteria In Solid Tumors 1.1 or Kaposi's sarcoma response criteria, which includes RECIST for visceral disease, or by Response Evaluation Criteria in Lymphoma for classical Hodgkin lymphoma [cHL]) and their corresponding 95% confidence intervals (calculated using exact binomial) will be reported separately for solid tumor and cHL according to treatment (combination therapy and single agent) using designated response criteria. Descriptive statistics will also be compiled for duration of response.
Time Frame: Up to 3 years
Population: Patients exposed to at least a single dose of study drug(s)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors | Dose Expansion Nivolumab 240 mg q2w and Ipilimumab 1 mg/kg q6w | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma
Number analyzed (Participants) | 5 | 8 | 7 | 4 | 23 | 20 | 9
Participants
  Complete Response | 0 | 0 | 0 | 1 | 0 | 2 | 2
  Partial Response | 2 | 0 | 0 | 1 | 7 | 4 | 5
  Objective Response (complete or partial response) | 2 | 0 | 0 | 2 | 7 | 6 | 7

5. Secondary Outcome: Immune Function, Defined as CD4 and CD8 Cell Counts at Baseline and at End of 46 Cycles of Treatment+ 6 Weeks
Description: Descriptive statistics will be generated to evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab, on immune function (CD4 and CD8 cells). Changes in CD4+ T-cell counts, CD8+ T-cell from baseline to end of 46 cycles of treatment+ 6 weeks visit were evaluated by Wilcoxon signed-rank test for paired data.
Time Frame: end of 46 cycles of treatment+ 6 weeks
Population: Enrolled participants who have data available for both baseline and end of 46 cycles of treatment+ 6 weeks visit
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors | Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 11 | 11 | 7
cells/mm3
  CD4+ T-cell counts at baseline | 322 [283 to 400] | 150 [115 to 152] | 563 [254 to 933] | 201 [106 to 203] | 412 [295 to 487] | 433 [232 to 594] | 319 [287 to 588]
  CD4+ T-cell counts at end of 46 cycles of treatment+ 6 weeks | 323 [240 to 565] | 125 [87 to 138] | 681 [308 to 899] | 177.5 [122 to 233] | 296 [203 to 427] | 422 [308 to 846] | 547 [237 to 661]
  CD8+ T-cell counts at baseline | 784 [778 to 791] | 380 [275 to 420] | 758 [657 to 789] | 311 [288 to 561] | 947 [348 to 1183] | 703 [514 to 1073] | 638 [302 to 1309]
  CD8+ T-cell counts at end of 46 cycles of treatment+ 6 weeks | 516 [476 to 1021] | 192 [161 to 260] | 737 [632 to 909] | 433 [198 to 668] | 584 [275 to 874] | 603 [551 to 1195] | 760 [424 to 1048]
Statistical Analysis 1: Comparison: Dose De-escalation Nivolumab 3mg/kg (Stratum 1); Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dose De-escalation Nivolumab 3 mg/kg (Stratum 2); Changes in CD4+ T-cell counts from baseline toend of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 0.6719, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1); Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 0.5000, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2); Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Dose Expansion Nivolumab 240 mg q2w in Solid Tumors; Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 0.1475, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg; Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 0.0420, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma; Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Dose De-escalation Nivolumab 3mg/kg (Stratum 1); Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 0.5000, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Dose De-escalation Nivolumab 3 mg/kg (Stratum 2); Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 0.1563, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) vs Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2); Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2); Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Dose Expansion Nivolumab 240 mg q2w in Solid Tumors; Changes in CD8+ T-cell counts from baseline to post-treatment last visit; Test type: Superiority; p = 0.2324, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg; Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 0.1016, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma; Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 0.8125, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Immune Function, Defined as CD4 and CD8 Cell Counts at Baseline and at End of 46 Cycles of Treatment+ 16 Weeks
Description: Descriptive statistics will be generated to evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab, on immune function (CD4 and CD8 cells). Changes in CD4+ T-cell counts, CD8+ T-cell from baseline to end of 46 cycles of treatment+ 16 weeks visit were evaluated by Wilcoxon signed-rank test for paired data.
Time Frame: end of 46 cycles of treatment+ 16 weeks
Population: Enrolled participants who have data available for both baseline and end of 46 cycles of treatment+ 16 weeks visit
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors | Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 11 | 8 | 5
cells/mm3
  CD4+ T-cell counts at baseline | 400 [284 to 443] | 152 [151 to 193] | 563 [254 to 933] | 106 [106 to 106] | 379 [295 to 720] | 391.5 [222 to 604.5] | 451 [319 to 588]
  CD4+ T-cell counts at end of 46 cycles of treatment+ 16 weeks | 270 [267 to 402] | 127 [60 to 199] | 692 [292 to 1122] | 197 [197 to 197] | 295 [242 to 707] | 441 [336.5 to 881] | 569 [400 to 577]
  CD8+ T-cell counts at baseline | 791 [784 to 1446] | 441 [420 to 462] | 758 [657 to 789] | 561 [561 to 561] | 1001.5 [828 to 1183] | 545 [473 to 707] | 1004 [638 to 1309]
  CD8+ T-cell counts at end of 46 cycles of treatment+ 16 weeks | 801 [499 to 1062] | 147 [139 to 251] | 956 [754 to 1019] | 616 [616 to 616] | 910 [293 to 1071] | 724.5 [563 to 879.5] | 1042 [679 to 1200]
Statistical Analysis 1: Comparison: Dose De-escalation Nivolumab 3mg/kg (Stratum 1); Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.5000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dose De-escalation Nivolumab 3 mg/kg (Stratum 2); Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.5000, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1); Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.2500, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2); Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Dose Expansion Nivolumab 240 mg q2w in Solid Tumors; Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.2061, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg; Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.0547, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma; Changes in CD4+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Dose De-escalation Nivolumab 3mg/kg (Stratum 1); Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.5000, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Dose De-escalation Nivolumab 3 mg/kg (Stratum 2); Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.500, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1); Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.500, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2); Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Dose Expansion Nivolumab 240 mg q2w in Solid Tumors; Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.0195, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg; Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.0234, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma; Changes in CD8+ T-cell counts from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.4375, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: HIV Viral Load at Baseline and at End of 46 Cycles of Treatment+ 6 Weeks
Description: Descriptive statistics will be generated to evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab, on HIV viral load. Changes in HIV viral load from baseline to end of 46 cycles of treatment+ 6 weeks visit were evaluated by Wilcoxon signed-rank test for paired data.
Time Frame: end of 46 cycles of treatment+ 6 weeks
Population: Enrolled participants who have data available for both baseline and end of 46 cycles of treatment+ 6 weeks visit
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors | Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma
Number analyzed (Participants) | 3 | 7 | 3 | 2 | 12 | 12 | 7
cells/mm3
  HIV viral load at baseline | 20 [10 to 20] | 10 [10 to 20] | 20 [10 to 20] | 19.5 [10 to 29] | 15 [10 to 20] | 20 [10 to 20] | 20 [10 to 47]
  HIV viral load at end of 46 cycles of treatment+ 6 weeks | 20 [10 to 20] | 10 [10 to 10] | 20 [20 to 36] | 40.5 [40 to 41] | 15 [10 to 20] | 20 [10 to 20] | 20 [10 to 40]
Statistical Analysis 1: Comparison: Dose De-escalation Nivolumab 3 mg/kg (Stratum 2); Changes in HIV viral load from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1); Changes in HIV viral load from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2); Test type: Superiority; p = 0.5000, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Dose Expansion Nivolumab 240 mg q2w in Solid Tumors; Changes in HIV viral load from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 0.5000, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg; Changes in HIV viral load from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 0.6250, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma; Changes in HIV viral load from baseline to end of 46 cycles of treatment+ 6 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: HIV Viral Load at Baseline and at End of 46 Cycles of Treatment+ 16 Weeks
Description: Descriptive statistics will be generated to evaluate the effects of single agent nivolumab, and the combination of ipilimumab and nivolumab, on HIV viral load. Changes in HIV viral load from baseline to end of 46 cycles of treatment+ 16 weeks visit were evaluated by Wilcoxon signed-rank test for paired data.
Time Frame: end of 46 cycles of treatment+16 weeks
Population: Enrolled participants who have data available for both baseline and end of 46 cycles of treatment+ 16 weeks visit
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors | Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 9 | 8 | 5
cells/mm3
  HIV viral load at baseline | 20 [10 to 20] | 10 [10 to 20] | 20 [10 to 20] | 10 [10 to 10] | 10 [10 to 20] | 20 [15 to 20] | 36 [20 to 47]
  HIV viral load at end of 46 cycles of treatment+ 16 weeks | 20 [10 to 20] | 10 [10 to 20] | 20 [10 to 60] | 10 [10 to 10] | 20 [10 to 20] | 20 [15 to 20] | 20 [20 to 30]
Statistical Analysis 1: Comparison: Dose Expansion Nivolumab 240 mg q2w in Solid Tumors; Changes in HIV viral load from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg; Changes in HIV viral load from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 0.7500, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma; Changes in HIV viral load from baseline to end of 46 cycles of treatment+ 16 weeks; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)

9. Other Pre Specified Outcome: Intratumor Immune Cells
Description: Will be assessed by immunohistochemistry. Descriptive statistics will be generated. Changes from pre-study to end of study will be explored using nonparametric Wilcoxon signed-rank test.
Time Frame: Up to 3 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Circulating Cytokine Markers
Description: Will be assessed by multiplex assay. Descriptive statistics will be generated. Changes from pre-study to end of study will be explored using nonparametric Wilcoxon signed-rank test.
Time Frame: Up to 3 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Herpesvirus Loads (Epstein-Barr Virus [EBV], Kaposi Sarcoma Herpes Virus [KSHV], Cytomegalovirus [CMV]) in Plasma
Description: Descriptive statistics will be generated. Changes from pre-study to end of study will be explored using nonparametric Wilcoxon signed-rank test.
Time Frame: Up to 3 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Latent Herpesvirus (EBV, KSHV, CMV) in Peripheral Blood Mononuclear Cell (PBMC)
Description: as for outcome 11
Time Frame: Up to 3 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Herpesvirus Specific CD8 and CD4 T Cells in PBMC
Description: as for outcome 11
Time Frame: Up to 3 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Viral Transcription in Tumor Biopsies (Kaposi Sarcoma Cases)
Description: as for outcome 11
Time Frame: Up to 3 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Human Papillomavirus Types in Anal Swabs (Anal Cancer Cases)
Description: as for outcome 11
Time Frame: Up to 3 years
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Latent HIV Loads in PBMC
Description: Will be assessed using outgrowth assay. Descriptive statistics will be generated. Changes from pre-study to end of study will be explored using nonparametric Wilcoxon signed-rank test.
Time Frame: Up to 3 years
Reporting Status: Not Posted

17. Other Pre Specified Outcome: HIV Reactive T Cells
Description: as for outcome 11
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants were followed for 16 weeks or 112 days (based on 5 half lives) after removal from study treatment, or until death, whichever occured first. Participants removed from study for unacceptable adverse event(s) were followed until resolution or stabilization of the adverse event.
Description: All adverse events, irrespective of their attribution have been included.
Arm/Group | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors | Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma
All-Cause Mortality (participants affected / at risk) | 0/6 | 3/9 | 1/7 | 2/4 | 5/24 | 1/20 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/6 | 6/9 | 3/7 | 3/4 | 9/24 | 6/20 | 2/9
Other Adverse Events (participants affected / at risk) | 5/6 | 8/9 | 6/7 | 4/4 | 22/24 | 20/20 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) (N=6) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) (N=9) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) (N=7) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2) (N=4) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors (N=24) | Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg (N=20) | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma (N=9)
CARDIAC ARREST (CARDIAC DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIAC DISORDERS - OTHER, SPECIFY (CARDIAC DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Cardiomyopathy
PERICARDIAL TAMPONADE (CARDIAC DISORDERS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADRENAL INSUFFICIENCY (ENDOCRINE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOTHYROIDISM (ENDOCRINE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASCITES (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHEA (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ORAL HEMORRHAGE (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEATH NOS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DISEASE PROGRESSION (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unspecified natural causes
HEPATIC FAILURE (HEPATOBILIARY DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — COVID-19
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — COVID-19 Infection
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Parainfluenza 3
LUNG INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH PUSTULAR (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (INFECTIONS AND INFESTATIONS) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0)
UPPER RESPIRATORY INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FRACTURE (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Post op neck swelling & dysphagia
ALANINE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
HYPONATREMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — bilateral temporomandibular joint dysfunction (TMJ) dislocation
PAIN IN EXTREMITY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Burkitt's Lymphoma
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Left eye biopsy consistent with Metastatic Squamous Cell carcinoma
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient's death likely attributed to progression of disease and died on 29 December 2017.
ENCEPHALOPATHY (NERVOUS SYSTEM DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (RENAL AND URINARY DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ASPIRATION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATELECTASIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Skin thickening rash
HYPOTENSION (VASCULAR DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose De-escalation Nivolumab 3mg/kg (Stratum 1) (N=6) | Dose De-escalation Nivolumab 3 mg/kg (Stratum 2) (N=9) | Dose De-escalation Nivolumab 240mg and Ipilimumab 1 mg/kg (Stratum 1) (N=7) | Dose De-escalation Nivolumab 240 mg and Ipilimumab 1mg/kg (Stratum 2) (N=4) | Dose Expansion Nivolumab 240 mg q2w in Solid Tumors (N=24) | Dose Expansion Nivolumab 240 mg and Ipilimumab 1 mg/kg (N=20) | Nivolumab 240 mg q2w in Classical Hodgkin Lymphoma (N=9)
ANEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (8) | 1 (2)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Swollen lymph node - left neck
SINUS BRADYCARDIA (CARDIAC DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (EAR AND LABYRINTH DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — left ear congestion
EAR PAIN (EAR AND LABYRINTH DISORDERS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHYROIDISM (ENDOCRINE DISORDERS) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
BLURRED VISION (EYE DISORDERS) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
DRY EYE (EYE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
EYE DISORDERS - OTHER, SPECIFY (EYE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Irritated, erythematous right eye probably due to foreign body
EYE DISORDERS - OTHER, SPECIFY (EYE DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — bilateral eye pressure
RETINAL VASCULAR DISORDER (EYE DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UVEITIS (EYE DISORDERS) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
ANAL HEMORRHAGE (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANAL PAIN (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOATING (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COLITIS (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (GASTROINTESTINAL DISORDERS) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
DENTAL CARIES (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHEA (GASTROINTESTINAL DISORDERS) | 4 (6) | 2 (3) | 4 (8) | 1 (1) | 3 (4) | 7 (12) | 3 (4)
DRY MOUTH (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPEPSIA (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
FLATULENCE (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Neck "Fullness"
GINGIVAL PAIN (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUCOSITIS ORAL (GASTROINTESTINAL DISORDERS) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (GASTROINTESTINAL DISORDERS) | 2 (2) | 2 (2) | 4 (8) | 2 (2) | 4 (5) | 5 (16) | 4 (6)
ORAL DYSESTHESIA (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL HEMORRHAGE (GASTROINTESTINAL DISORDERS) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL PAIN (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
RECTAL FISTULA (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOOTHACHE (GASTROINTESTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (GASTROINTESTINAL DISORDERS) | 2 (2) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 4 (12) | 2 (2)
CHILLS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (1)
EDEMA FACE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EDEMA LIMBS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 5 (7) | 1 (1)
FATIGUE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 3 (7) | 4 (5) | 3 (6) | 3 (3) | 8 (9) | 10 (17) | 3 (5)
FEVER (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 1 (1)
FLU LIKE SYMPTOMS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GAIT DISTURBANCE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NON-CARDIAC CHEST PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 6 (12) | 2 (2)
ANORECTAL INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLADDER INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHIAL INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Human Corona Virus (HKU1) Infection
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — TB-Latent
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — norovirus infection
LUNG INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PAPULOPUSTULAR RASH (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
SKIN INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (2)
THRUSH (INFECTIONS AND INFESTATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOOTH INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
BRUISING (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
ALKALINE PHOSPHATASE INCREASED (INVESTIGATIONS) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (7)
BLOOD LACTATE DEHYDROGENASE INCREASED (INVESTIGATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
CD4 LYMPHOCYTES DECREASED (INVESTIGATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
CREATININE INCREASED (INVESTIGATIONS) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (7) | 2 (3)
INVESTIGATIONS - OTHER, SPECIFY (INVESTIGATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Elevated C-reactive protein, free kappa light chains, free lambda light chains, and IgM
INVESTIGATIONS - OTHER, SPECIFY (INVESTIGATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Phosphorus decreased
INVESTIGATIONS - OTHER, SPECIFY (INVESTIGATIONS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — UREA NITROGEN INCREASED
LIPASE INCREASED (INVESTIGATIONS) | 2 (10) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
LYMPHOCYTE COUNT DECREASED (INVESTIGATIONS) | 2 (9) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9)
NEUTROPHIL COUNT DECREASED (INVESTIGATIONS) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (7)
PLATELET COUNT DECREASED (INVESTIGATIONS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
SERUM AMYLASE INCREASED (INVESTIGATIONS) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (11) | 2 (5) | 1 (3)
THYROID STIMULATING HORMONE INCREASED (INVESTIGATIONS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WEIGHT GAIN (INVESTIGATIONS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
WEIGHT LOSS (INVESTIGATIONS) | 1 (4) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL DECREASED (INVESTIGATIONS) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (9) | 0 (0) | 5 (11)
ANOREXIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 2 (3) | 2 (3) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
DEHYDRATION (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKALEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
HYPERNATREMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOALBUMINEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (5)
HYPOCALCEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
HYPOGLYCEMIA (METABOLISM AND NUTRITION DISORDERS) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
HYPONATREMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (7) | 3 (3)
HYPOPHOSPHATEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 2 (3)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Food aversion
ARTHRALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (10) | 3 (3) | 0 (0)
ARTHRITIS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
FLANK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUSCLE CRAMP (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
NECK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
TUMOR PAIN (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
DIZZINESS (NERVOUS SYSTEM DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1)
DYSGEUSIA (NERVOUS SYSTEM DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (NERVOUS SYSTEM DISORDERS) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 3 (5) | 6 (7) | 1 (3)
LETHARGY (NERVOUS SYSTEM DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARESTHESIA (NERVOUS SYSTEM DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (NERVOUS SYSTEM DISORDERS) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
PRESYNCOPE (NERVOUS SYSTEM DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (NERVOUS SYSTEM DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
VASOVAGAL REACTION (NERVOUS SYSTEM DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (PSYCHIATRIC DISORDERS) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
INSOMNIA (PSYCHIATRIC DISORDERS) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PSYCHIATRIC DISORDERS - OTHER, SPECIFY (PSYCHIATRIC DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — panic attacks
CHRONIC KIDNEY DISEASE (RENAL AND URINARY DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (RENAL AND URINARY DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (RENAL AND URINARY DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — cortisol decreased
URINARY FREQUENCY (RENAL AND URINARY DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (RENAL AND URINARY DISORDERS) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY URGENCY (RENAL AND URINARY DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENITAL EDEMA (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VAGINAL HEMORRHAGE (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHIAL OBSTRUCTION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (2) | 1 (1) | 1 (3) | 3 (4) | 7 (8) | 6 (7) | 4 (8)
DYSPNEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 7 (9) | 1 (1)
EPISTAXIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HOARSENESS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
NASAL CONGESTION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (3)
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POSTNASAL DRIP (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
RHINORRHEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
SNEEZING (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SORE THROAT (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ALOPECIA (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRY SKIN (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HYPERHIDROSIS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERTRICHOSIS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 6 (7) | 1 (2)
RASH ACNEIFORM (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 5 (9) | 4 (7) | 3 (4)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Lower Back Nodule
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Rash
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — papule - buttock
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (SURGICAL AND MEDICAL PROCEDURES) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Tooth Extraction
HOT FLASHES (VASCULAR DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hot Flashes
HYPERTENSION (VASCULAR DISORDERS) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 6 (15) | 8 (17) | 1 (1)
HYPOTENSION (VASCULAR DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
THROMBOEMBOLIC EVENT (VASCULAR DISORDERS) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT02408861/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT02408861/ICF_001.pdf